CLINICAL TRIAL: NCT02283866
Title: Bispectral Index-Guided Versus Fixed Dose Administration of Desflurane During Balanced Anesthesia With Remifentanil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CWJung_BA
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Stabilizing Hypnotic Depth and Vital Sign During Balanced Anesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Administering desflurane according to the patient's BIS value (Experimental): The anesthesiologist administers the volatile anesthetic desflurane to set the patient's BIS value at 50 during balanced anesthesia, and titrate the remifentanil dose to set the patient's systolic arterial blood pressure between 100-140mmHg.
  Interventions: Drug: Administering desflurane according to the patient's BIS value
- Administering desflurane at 1 MAC (Experimental): The anesthesiologist administers the volatile anesthetic desflurane at 1 MAC during balanced anesthesia, and titrate the remifentanil dose to set the patient's systolic arterial blood pressure between 100-140mmHg.
  Interventions: Drug: Administering desflurane at 1 MAC

INTERVENTIONS:
Drug: Administering desflurane according to the patient's BIS value — Administering desflurane according to the patient's BIS value
  Arms: Administering desflurane according to the patient's BIS value
Drug: Administering desflurane at 1 MAC — Administering desflurane at 1 MAC
  Arms: Administering desflurane at 1 MAC

SUMMARY:
Balanced anesthesia combining volatile anesthetics and opioids is commonly used in modern anesthesia. The purpose of this study is to compare two methods of administering desflurane, an volatile anesthetic during balanced anesthesia. The investigators hypothesized that administering desflurane at 1 MAC (minimum alveolar concentration) during balanced anesthesia will be more beneficial in terms of stability of the patient's vital signs and hypnotic depth than administering desflurane according to the patient's BIS (bispectral index) value.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for operation under balanced anesthesia using desflurane and remifentanil

Exclusion Criteria:

* Refusal of consent
* General anesthesia with agents other than desflurane and remifentanil
* Patients with allergy to neuromuscular blocker, volatile anesthetics, opioids
* History of malignant hyperthermia
* Patients taking CNS stimulants
* Chronic alcohol abuser
* Patients with severe depressed left ventricular function, EF < 30%
* Patients with convulsive disorders
* ASA class IV, V, VI
* Patients with systolic arterial blood pressure lower than 90mmHg before surgery
* Patients needing inotropic infusion during surgery
* Anesthesia time less than 30 minutes

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The difference of 'wobble' value of the patients' BIS value between the two groups | Every second from 10 minutes after skin incision to 10 minutes before surgery end.
  'Wobble' is a variable that can measure the performance measurement of a pharmacokinetic model, or the reaction of the patient to a drug. We can calculate the performance error from the target of the therapy and the actual measured value, and derive the wobble by a specific formulas, which are described below.
  PE=(BISmeasured-BIStargeted)x100/BIStargeted MDPEi = median{PEij, j=1,…,Ni} MDAPEi = median{|PEij|, j=1,…,Ni} Wobblei = median{|PEij-MDPEi|, j=1,…,Ni} Divergence = slope{|PEij|, j=1,…,Ni}

SECONDARY OUTCOMES:
The difference of 'wobble' value of the patients' systolic arterial blood pressure value between the two groups | Every 2.5 minutes from 10 minutes after skin incision to 10 minutes before surgery end
  Described above

OTHER OUTCOMES:
Eye opening time to prodding after stopping of anesthetics. | 1 min,2 min,3 min, 4min, 5min, 6min, 7min, 8min, 9min, 10min after stopping injection of anesthetics

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yang SM, Jung YS, Jung CW, Kim WH, Yoon SB, Lee HC. Comparison of bispectral index-guided and fixed-gas concentration techniques in desflurane and remifentanil anesthesia: A randomized controlled trial. PLoS One. 2020 Nov 5;15(11):e0241828. doi: 10.1371/journal.pone.0241828. eCollection 2020. PMID 33152029